CLINICAL TRIAL: NCT04365673
Title: Comparing the Predictive Strength of the LACE+ Index With the MedWise Rise Score on Hospital Readmission Rates: a Non-inferiority Observational Study
Brief Title: LACE+ and MRS Score Readmission Rate Assessment
Status: Terminated | Type: Observational
Why Stopped: Terminated: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention. Lack of data to demonstrate sufficient power.
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: TRHC_RD_LACEMRS_2020
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Hospitalism
Keywords: LACE; medication risk score

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Readmitted: Patients that were readmitted within 30 days post hospital discharge
  Interventions: Other: Pharmacist transition of care consultation
- Not readmitted: Patients that were not readmitted within 30 days post hospital discharge
  Interventions: Other: Pharmacist transition of care consultation

INTERVENTIONS:
Other: Pharmacist transition of care consultation — Pharmacist-delivered comprehensive medication review

SUMMARY:
A study to demonstrate that the LACE+ score in non-inferior to the medication risk score when predicting 30-day readmission post hospital discharge.

DETAILED DESCRIPTION:
The objective of this study is evaluate a program that provides transition of care services to a local Tucson hospital involving activities designed to reduce 30 day post hospital discharge readmission rates. The organization has had a fee for service contract with this hospital since 2017 to provide pharmacist delivered transition of care services. The organization collects internal tracking outcome data as part of the contract deliverable and is required to report it to the hospital once per month. The investigators look to assess LACE+ and medication risk scores to learn if there is an association with the 30 day post hospital discharge readmission rate post pharmacist intervention. The outcomes will not be generalizable and will be reported back to the hospital client to demonstrate value added.

ELIGIBILITY:
Inclusion Criteria:

* Those referred to receive transition of care services between January 2018 to December 2019 and were discharged on 10 or more medications.

Exclusion Criteria:

* 89 years or older

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Information will be collected from an internal data collection excel used to provide monthly outcome intervention reports to the local Tucson hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Readmission | 2018 - 2019
  Readmission within 30-days post hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bingham, PharmD, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Tabula Rasa HealthCare, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided